CLINICAL TRIAL: NCT05659173
Title: Association of Vitamin D Deficiency With Selected Vitamin D Receptor (VDR) Gene Polymorphism in Gestational Hypertension Among Malaysian Women: A Prospective Genetic Biomarker for Early Intervention Strategy
Brief Title: Vitamin D Deficiency With Selected Vitamin D Receptor Gene Polymorphism in Gestational Hypertension
Status: Active, not recruiting | Type: Observational
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Ministry of Higher Education, Malaysia (Other)
Responsible Party: Principal Investigator, Nurul Iftida Binti Basri, Dr, Universiti Putra Malaysia
Other Study IDs: FRGS/1/2022/SKK01/UPM/02/1
Record Dates: First submitted 2022-11-06; First posted 2022-12-21 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Hypertensive Disorder of Pregnancy; Vitamin D Deficiency
MeSH Terms: conditions — Toxemia; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood for vitamin D level and genomic DNA decsription
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1- normotensive women: Women with vitamin D deficiency and normotensive during pregnancy
  Interventions: Diagnostic Test: Blood taking
- 2- women with hypertensive disorder in pregnancy: Women with Vitamin D deficiency and hypertensive disorder in pregnancy
  Interventions: Diagnostic Test: Blood taking

INTERVENTIONS:
Diagnostic Test: Blood taking — Blood test for vitamin D level and DNA extraction for VDR gene polymorphism

SUMMARY:
This study aim to look into the prevalence of Vitamin D deficiency among Malaysian pregnant women and its associated risk factors. Subsequently, vitamin D deficient women with and without gestational hypertension will be investigated for their genetic variation to look for the association of VDR genetic variation and hypertensive disorders in pregnancy.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy account for approximately 14% of maternal mortality globally and is the fourth leading cause of maternal mortality in Malaysia. Despite this, the mechanisms and pathogenesis are still unknown. Vitamin D deficiency (hypovitaminosis vitamin D) has been shown to be one of the causes of gestational hypertension(GH).

Several populations have observed the association of single nucleotide polymorphisms (SNPs) of vitamin D receptor (VDR) to vitamin D deficiency among pregnancy complications, including GH. Alarming cases of hypovitaminosis D in sunny areas including Malaysia, highly imply the need to understand the genetic factor. Hence, genotyping VDR variants among pregnant women is essential for early vitamin D supplementation strategy. To investigators knowledge, there has been no published study conducted among Malaysian population on the association of VDR genetic variation and GH. Therefore, this study aim to investigate the prevalence of vitamin D deficiency and its association of VDR SNPs to the development of GH among Malaysian pregnant mothers, with the main focus on Malays, representing the largest ethnic in Malaysia.

The prevalence will be determined through a cross-sectional study involving 363 pregnant women recruited in Hospital Pengajar UPM (HPUPM) and Hospital Serdang, Selangor. Relevant socio-demographic, clinical and anthropometric data will be collected using structured interviewer-administered questionnaire. Blood specimens for the analysis of vitamin D will be done. The association will be determined in a case-control study involving 180 pregnant women who fulfilled the criteria, recruited from phase 1 study. Their blood will be further analysed for the variants of the VDR gene [(BsmI(rs1544410), FokI(rs2228570), TaqI(rs731236)] to look for the association.

This study expected to provide more evidence for early personalised intervention of vitamin D supplementation due to anticipated individual genetic variability. This antenatal care programme will reduce the government expenditures, reduce maternal and fetal morbidity and mortality while strengthening Malaysia's healthcare system.

ELIGIBILITY:
Inclusion Criteria:

1. Malay pregnant women with gestational age between 20 weeks till 42 weeks. (The gestational age will be determined from the first day of the last menstrual cycle or measurement of fetal crown rump length)
2. Malay pregnant women with viable pregnancy with or without pregnancy induced hypertension or its complications (pre-eclampsia, eclampsia, HELLP syndrome etc).
3. Literate in either English or Malay languages.
4. Agreement to follow-up till delivery and provision of written informed consent.

Exclusion Criteria:

1. Non-viable pregnancy at the time of recruitment.
2. Women already on vitamin D supplements or any other drugs that can interfere with vitamin D absorption or metabolism at the time of recruitment.
3. Women with chronic hypertension diagnosed prior to pregnancy.
4. Pregnant women with any other chronic disease that is known to affect vitamin D such as, autoimmune disease and any malignancy

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All Malaysia pregnant women attending Obstetrics and Gynaecology Department of Hospital Pengajar UPM(HPUPM) and Hospital Serdang who fulfilled the criteria will be recruited.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of vitamin D deficiency | 1 year
  To determine the prevalence of Vitamin D deficiency among Malaysian pregnant mothers
Risk factors of vitamin D deficiency | 1 year
  To determine the associated risk factors of vitamin D deficiency among Malaysian pregnant mothers-weight, height and BMI will be measured in kg/m2.
Risk factors of vitamin D deficiency | 1 year
  To determine the associated risk factors of vitamin D deficiency among Malaysian pregnant mothers-duration of sun exposure in a week, measured in hours
Risk factors of vitamin D deficiency | 1 year
  To determine the associated risk factors of vitamin D deficiency among Malaysian pregnant mothers-intake of food rich in vitamin D, measured in serving number per week
VDR allele and genotype | 1 year
  To understand and associate distributions of VDR allele and genotype with vitamin D deficiency among Malay pregnant mothers
VDR-combined genotypes and gestational hypertension | 6 months
  To associate VDR-combined genotypes with the risk to develop gestational hypertension in vitamin D deficient Malay pregnant women

CONTACTS AND LOCATIONS:
Overall Officials: Nurul I Basri, MbChb, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Hospital Pengajar UPM, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ibrahim Y, Basri NI, Nordin N, Mohd Jamil AA. Vitamin D Deficiency and Its Association With Vitamin D Receptor Gene Variants Among Malaysian Women With Hypertensive Disorders in Pregnancy: Protocol for a Nutrigenomics Study. JMIR Res Protoc. 2024 Mar 26;13:e53722. doi: 10.2196/53722. PMID 38530345